CLINICAL TRIAL: NCT07013500
Title: Comparison of Gasserian Ganglion Conventional Radiofrequency and Peripheral Pulsed Radiofrequency in Trigeminal Neuralgia
Brief Title: Comparison of Two Types of Radiofrequency Treatment for Trigeminal Neuralgia
Acronym: TN-RFA-MEU25
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mesut Bakır (Other)
Responsible Party: Sponsor-Investigator, Mesut Bakır, Assoc. Prof. Dr. Mesut Bakır, Mersin University, Department of Algology, Mersin University
Organization: Mersin University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MERSINALG-TN-RFA-2025
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Trigeminal Neuralgia; Tic Douloureux; Neuropathic Facial Pain
Keywords: Trigeminal Neuralgia; Radiofrequency Ablation; Pulsed Radiofrequency; Gasserian Ganglion; Neuropathic Pain
MeSH Terms: conditions — Trigeminal Neuralgia; Neuralgia

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study.
Masking Description: Participants and investigators know which intervention is being received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Radiofrequency (Active Comparator): Patients in this group received conventional thermal radiofrequency (RFA) treatment targeting the Gasserian ganglion. The procedure was performed under fluoroscopic guidance using standard techniques. Lesioning was applied at 70-75°C for 60-90 seconds after correct positioning was confirmed with sensory and motor stimulation.
  Interventions: Procedure: Conventional Gasserian Ganglion Radiofrequency
- Peripheral Pulsed Radiofrequency (Experimental): Patients in this group received pulsed radiofrequency (PRF) applied peripherally to the affected branch of the trigeminal nerve (V1, V2, or V3), depending on the pain distribution. The procedure was performed under fluoroscopic guidance. PRF was applied at 42°C for two cycles of 120 seconds.
  Interventions: Procedure: Peripheral Pulsed Radiofrequency

INTERVENTIONS:
Procedure: Conventional Gasserian Ganglion Radiofrequency — Conventional RFA was performed at the Gasserian ganglion under fluoroscopic guidance with thermal lesioning at 70-75°C for up to 90 seconds. Sensory and motor stimulation were used to verify needle placement.
  Arms: Conventional Radiofrequency
Procedure: Peripheral Pulsed Radiofrequency — PRF was applied to the peripheral branch of the trigeminal nerve at 42°C for two cycles of 120 seconds using fluoroscopic guidance. This technique was preferred in our clinic to avoid thermal complications such as hypoesthesia or motor dysfunction.
  Arms: Peripheral Pulsed Radiofrequency

SUMMARY:
Trigeminal neuralgia (TN) is a chronic pain condition that affects the face, often causing sharp, electric shock-like pain in areas served by the trigeminal nerve. When medications are no longer effective, interventional procedures such as radiofrequency ablation (RFA) may be used. This retrospective study compares two different RFA techniques in patients with classical TN: (1) conventional thermal RFA applied to the Gasserian ganglion, and (2) pulsed RFA applied peripherally to the nerve branches.

The purpose of the study is to evaluate pain relief, patient satisfaction, and complication rates between these two commonly used techniques. A total of 60 patients aged 55-80 years, who were treated at the Mersin University Pain Clinic between January 2015 and June 2025, were included. The study uses clinical records and follow-up data to assess outcomes at 6 months post-procedure.

This study aims to provide clinicians with more evidence to guide the selection of safer and more effective treatments for trigeminal neuralgia, with the goal of improving patients' quality of life and reducing treatment-related side effects.

DETAILED DESCRIPTION:
Trigeminal neuralgia (TN) is a debilitating neuropathic condition characterized by recurrent episodes of severe, lancinating facial pain in the distribution of one or more branches of the trigeminal nerve. Although most patients initially respond to medical therapy such as carbamazepine or oxcarbazepine, a subset remains refractory and requires interventional treatment.

Radiofrequency ablation (RFA) has been widely used in the management of refractory TN, especially conventional thermal RFA targeting the Gasserian ganglion. While this approach offers substantial pain relief, it may lead to complications such as facial numbness, dysesthesia, or weakness due to irreversible nerve damage. As an alternative, pulsed RFA (PRF) offers neuromodulation without causing structural nerve injury and is often preferred for peripheral branch interventions.

This retrospective cohort study aims to compare the effectiveness and safety of two RFA techniques in patients with classical TN:

Group A: Conventional RFA applied to the Gasserian ganglion

Group B: Pulsed RFA applied peripherally to the affected branch (V1, V2, or V3)

Patients were selected from the records of the Pain Clinic of Mersin University Faculty of Medicine between January 1, 2015, and June 1, 2025. A total of 60 patients aged 55-80 years, who had been diagnosed with classical TN (per ICHD-3 criteria), were included. All patients had failed medical management for at least 6 months and underwent either of the RFA techniques described above. Patients with secondary TN, prior craniofacial surgery, or missing follow-up data were excluded.

PRF was specifically chosen for peripheral interventions in our clinic to avoid thermal-related complications. PRF was applied at 42°C for two cycles of 120 seconds. Thermal RFA was applied with standard lesioning parameters following contrast-confirmed Gasserian ganglion targeting.

Outcome measures included:

Primary: Pain relief measured using a numerical rating scale (NRS) at baseline and 6 months post-procedure

Secondary: Patient satisfaction (5-point Likert scale), rate of complications, and recurrence of pain requiring reintervention

All procedures were performed under fluoroscopic guidance by experienced pain specialists. Data was extracted from electronic records and procedure reports. Statistical comparisons will be made using appropriate parametric or non-parametric tests based on data distribution.

This study seeks to contribute real-world evidence to guide clinicians in selecting safer, more effective RFA strategies for managing TN, particularly in patients at risk for complications or those preferring less invasive approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 55 and 80 years with a diagnosis of classical trigeminal neuralgia according to the International Classification of Headache Disorders, 3rd edition (ICHD-3). Patients must have experienced pain refractory to medical management for at least 6 months and have complete clinical and procedural records available, including follow-up data for a minimum of 6 months.

Exclusion Criteria:

* Patients with secondary trigeminal neuralgia due to structural causes such as multiple sclerosis or tumors, those with a history of prior craniofacial surgery or neuroablative procedures, patients lacking sufficient follow-up data, and those with contraindications to sedation or with uncontrolled systemic comorbidities are excluded from the study.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Reduction | Baseline and 6 months after intervention
  Change in pain intensity score measured on the Numerical Rating Scale (NRS) from baseline to 6 months post-procedure.

SECONDARY OUTCOMES:
Patient Satisfaction Score | 6 months post-procedure
  Patient-reported satisfaction with the intervention, measured using a 5-point Likert scale at the 6-month follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mesut Bakır, Assoc. Prof, Principal Investigator — Mersin University Faculty of Medicine, Pain Clinic
Locations (1):
- Mersin University Faculty of Medicine, Department of Algology, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes will be shared upon reasonable request. Data will be available after publication and can be requested by contacting the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data and selected supporting documents will be available upon request beginning 6 months after publication. Data will remain available for 5 years.
Access Criteria: Researchers affiliated with academic institutions may request access to anonymized individual participant data and related documents for non-commercial research. Requests must include a brief study proposal and will be reviewed by the principal investigator. Data will be shared via institutional email upon approval.

REFERENCES:
- [Background] Chua NH, Vissers KC, Sluijter ME. Pulsed radiofrequency treatment in interventional pain management: mechanisms and potential indications-a review. Acta Neurochir (Wien). 2011 Apr;153(4):763-71. doi: 10.1007/s00701-010-0881-5. Epub 2010 Nov 30. PMID 21116663
- [Derived] Bakir M, Turkyilmaz GG, Teker N, Yavuz K, Ilcan B, Rumeli S. Comparison of Gasserian ganglion conventional radiofrequency ablation and peripheral nerve pulsed radiofrequency in trigeminal neuralgia: a retrospective cohort study. J Oral Facial Pain Headache. 2026 Jan;40(1):119-126. doi: 10.22514/jofph.2025.063. Epub 2026 Jan 12. PMID 41607329